CLINICAL TRIAL: NCT03779893
Title: Clinical Evaluation of Bioactive Resin Based Pits & Fissures Sealants Versus Conventional Resin Based Pits & Fissures Sealants in Caries Susceptible Fissures in Permanent Molars: A Randomized Controlled Trial
Brief Title: Clinical Evaluation of Bioactive Resin Sealants vs Conventional Sealants in Permanent Molars
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fathi Abdelsalam, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14011989
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): Conventional resin based Pits & fissures sealant 3M™ Clinpro™ Sealant is administrated
  Interventions: Combination Product: 3M™ Clinpro™ Sealant.
- bioactive group (Experimental): Bioactive Pits & fissures sealant BioCoat® by Premier®.
  Interventions: Combination Product: BioCoat® by Premier®.

INTERVENTIONS:
Combination Product: BioCoat® by Premier®. — Bioactive pits and fissure sealant
  Arms: bioactive group
Combination Product: 3M™ Clinpro™ Sealant. — conventional pits and fissure sealant
  Arms: conventional group

SUMMARY:
This study will be conducted to evaluate the performance; in terms of retention and caries inhibition; of the newly introduced bioactive resin based pits and fissure sealant versus conventional resin based pits and fissure sealant in caries susceptible fissures in posterior molars in patients at risk of caries. Evaluation will be done by visual tactile examination & VistaCAM.

DETAILED DESCRIPTION:
In the investigator's study the comparator material will be BioCoat® by Premier® ; new bioactive resin pits and fissures sealant featuring SmartCap™ Technology. SmartCap™ Technology utilizes patented semi-permeable resin microcapsules. In BioCoat, the rechargeable SmartCap microcapsules are filled with ionic solutions of fluoride, calcium and phosphate, which diffuse in and out of the sealant. Greater fluoride uptake in the presence of calcium and phosphate ions is assumed.

With limited evidence based information in literature about using bioactive fissure sealants in susceptible fissures , it was found beneficial to evaluate the newly introduced material using a randomized controlled trial to test the null hypothesis that bioactive resin pits and fissure sealant will have the same clinical performance as conventional resin based pits and fissure sealant in susceptible fissures.

ELIGIBILITY:
Inclusion Criteria of participants:

* Patients with bilateral caries susceptible fissures in molars showing no signs of caries.
* 19 - 40 years.
* Males or Females.
* Co-operative patients approving to participate in the trial.

Exclusion criteria of participants:

* Patients younger than 19 years old or older than 40 years old.
* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Allergic history concerning methacrylate.
* Rampant caries.
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of severe bruxism, clenching, or tempromandibular joint disorders.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Retention of sealant | one year
  rate of sealant loss

SECONDARY OUTCOMES:
Caries incidence | one year
  rate of caries initiation

IPD SHARING:
Plan to Share IPD: No